CLINICAL TRIAL: NCT00708500
Title: A Phase 3 Safety and Efficacy Study of Boceprevir in Subjects With Chronic Hepatitis C Genotype 1 Who Failed Prior Treatment With Peginterferon/Ribavirin
Brief Title: Boceprevir in Subjects With Chronic Hepatitis C Genotype 1 Who Failed Prior Treatment With Peginterferon/Ribavirin (Study P05101AM3)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05101; 2007-005151-42
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
Keywords: Treatment failure
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo+PEG2b+RBV, x 44 weeks (Placebo Comparator): Participants in Arm 1 (control) received pegylated interferon alfa 2b (PegIntron, PEG2b) + Ribavirin (RBV) (weight-based dosing [WBD]) for 4 weeks followed by boceprevir placebo + PEG2b + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
  Interventions: Biological: Pegylated interferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908); Drug: Boceprevir placebo
- Boceprevir+PEG2b+RBV, Response Guided Therapy (Experimental): Participants in Arm 2 (experimental) were assigned either a 36-week or 48-week course of therapy based on their HCV-RNA status at Treatment Week 8.
  PEG2b + RBV (WBD) for 4 weeks followed by boceprevir + PEG2b + RBV (WBD) for 32 weeks, then:
  * 36-week regimen: Participants who have undetectable HCV-RNA at Treatment Week 8 discontinue treatment and enter 36 weeks of post treatment follow-up.
  * 48-week regimen: Participants who have detectable HCV-RNA at Treatment Week 8 are assigned an additional 12 weeks of therapy, followed by 24 weeks of post treatment follow-up. Placebo replaces boceprevir for the remaining 12 weeks of therapy, and this switch will occur in a blinded fashion.
  Interventions: Drug: Boceprevir (SCH 503034); Biological: Pegylated interferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908); Drug: Boceprevir placebo
- Boceprevir+PEG2b+RBV, x 44 weeks (Experimental): Participants in Arm 3 (experimental) received PEG2b + RBV (WBD) for 4 weeks followed by boceprevir + PEG2b + RBV (WBD) for 44 weeks with 24 weeks post-treatment follow-up.
  Interventions: Drug: Boceprevir (SCH 503034); Biological: Pegylated interferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908)

INTERVENTIONS:
Drug: Boceprevir (SCH 503034) — Boceprevir, 200 mg capsules, 800 mg TID PO
  Arms: Boceprevir+PEG2b+RBV, Response Guided Therapy; Boceprevir+PEG2b+RBV, x 44 weeks
Biological: Pegylated interferon alfa-2b (SCH 54031) — PEG2b 1.5 μg/kg/week subcutaneously (SC)
  Other Names: PegIntron; PEG2b
Drug: Ribavirin (SCH 18908) — Ribavirin WBD 600 mg/day to 1400 mg/day by mouth (PO) divided twice daily (BID).
  Other Names: Rebetol; RBV
Drug: Boceprevir placebo — Boceprevir placebo, 200 mg capsules, 800 mg three times daily (TID) PO.
  Arms: Boceprevir+PEG2b+RBV, Response Guided Therapy; Placebo+PEG2b+RBV, x 44 weeks

SUMMARY:
This study involves treatment with boceprevir or placebo in combination with pegylated interferon alfa-2b (PegIntron, PEG2b) + Ribavirin (RBV) (weight-based dosing [WBD]) in adult subjects with chronic hepatitis C (CHC) genotype 1 who demonstrated interferon responsiveness (a decrease in hepatitis C virus RNA [HCV-RNA] viral load >=2 log10 by Week 12 or undetectable HCV-RNA at end of treatment) but who failed to achieve sustained virologic response (SVR) on prior treatment with any combination therapy of peginterferon alpha and RBV. This trial includes three arms, one control arm (PEG2b + RBV for 48 weeks) and two experimental arms (PEG2b + RBV + boceprevir). One of the experimental arms, Arm 3, consists of treatment with all three drugs for 44 weeks after the lead-in. The other experimental arm, Arm 2, consists of all three drugs for 32 weeks after the lead-in. Participants in Arm 2 who were undetectable for HCV-RNA at Treatment Week 8 will complete treatment at that point. Those who were not undetectable for HCV-RNA at Treatment Week 8 will receive an additional 12 weeks of PEG2b + RBV + boceprevir placebo. It is hypothesized that the addition of a third active anti-HCV drug may lead to more rapid viral response than therapy with two drugs, and therefore, the addition of boceprevir to PEG2b plus RBV therapy after a 4-week lead-in period may allow for both increased rates of SVR and shorter treatment durations (in some populations) than treatment with peginterferon plus RBV alone.

ELIGIBILITY:
Inclusion Criteria:

* Qualifying regimen defined as pegylated interferon alfa-2a plus ribavirin or pegylated interferon alfa-2b plus ribavirin for a minimum of 12 weeks.
* During qualifying regimen, participants must have either a documented undetectable HCV-RNA within 30 days of end of treatment (EOT) and a subsequent detectable HCV-RNA during follow-up or a documented decline in HCV-RNA by >=2 log10 by Treatment Week 12
* Previously documented CHC genotype 1 infection.
* Liver biopsy with histology consistent with CHC and no other etiology.
* Participants with bridging fibrosis or cirrhosis must have an ultrasound within 6 months of the Screening Visit (or between Screening and Day 1) with no findings suspicious for hepatocellular carcinoma (HCC).
* Participants participating in Schering-Plough Research Institute (SPRI) maintenance protocols P02570 (NCT00049842) or P02569 (NCT00048724) must have completed the study to be eligible for this protocol.
* Participants must be >=18 years of age.
* Participants must weigh between 40 kg and 125 kg.
* Participants and participant's partner(s) must each agree to use acceptable methods of contraception for at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations.
* Participants must be willing to give written informed consent.

Exclusion Criteria:

* Coinfection with the human immunodeficiency virus (HIV) or hepatitis B virus (Hepatitis B Surface Antigen [HBsAg] positive).
* Discontinuation of previous interferon or ribavirin regimen for an adverse event (AE) considered by the investigator to be possibly or probably related to ribavirin and/or interferon.
* Treatment with ribavirin within 90 days and any interferon-alpha within 1 month of Screening.
* Treatment for hepatitis C with any investigational medication. Prior treatment with herbal remedies with known hepatotoxicity.
* Treatment with any investigational drug within 30 days of the randomization visit.
* Participation in any other clinical trial within 30 days of randomization or intention to participate in another clinical trial.
* Evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy.
* Diabetic and/or hypertensive participants with clinically significant ocular examination findings.
* Pre-existing psychiatric conditions.
* Clinical diagnosis of substance abuse of the specified drugs within the specified timeframes
* Any known pre-existing medical condition that could interfere with the participant's participation in and completion of the study.
* Evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years (except adequately treated carcinoma in situ and basal cell carcinoma of the skin). Participants under evaluation for malignancy are not eligible.
* Participants who are pregnant or nursing. Participants who intend to become pregnant during the study period. Male participants with partners who are, or intend to become, pregnant during the study period.
* Any other condition which, in the opinion of a physician, would make the participant unsuitable for enrollment or could interfere with the participant participating in and completing the study.
* Participants who are part of the site personnel directly involved with this study.
* Participants who are family members of the investigational study staff.
* Participants who had life-threatening serious adverse event (SAE) during screening period.
* Protocol-specified hematologic, biochemical, and serologic criteria: Hemoglobin <12 g/dL for females and <13 g/dL for males; Neutrophils <1500/mm^3 (Blacks: <1200/mm^3); Platelets <100,000/mm^3; Direct bilirubin >1.5 x upper limit of normal (ULN).
* Serum albumin <lower limit of normal (LLN)
* Thyroid-stimulating hormone (TSH) >1.2 x ULN or <0.8 x LLN of laboratory reference range, with certain exceptions.
* Serum creatinine >ULN of the laboratory reference.
* Protocol-specified serum glucose concentrations.
* Protocol-specified alpha fetoprotein range.
* Prothrombin Time/Partial Thromboplastin Time (PT/PTT) values >10% above laboratory reference range.
* Anti-nuclear antibodies (ANA) >1:320.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Poordad F, Bronowicki JP, Gordon SC, Zeuzem S, Jacobson IM, Sulkowski MS, Poynard T, Morgan TR, Molony C, Pedicone LD, Sings HL, Burroughs MH, Sniukiene V, Boparai N, Goteti VS, Brass CA, Albrecht JK, Bacon BR; SPRINT-2 and RESPOND-2 Investigators. Factors that predict response of patients with hepatitis C virus infection to boceprevir. Gastroenterology. 2012 Sep;143(3):608-618.e5. doi: 10.1053/j.gastro.2012.05.011. Epub 2012 May 21. PMID 22626609
- [Derived] Bacon BR, Gordon SC, Lawitz E, Marcellin P, Vierling JM, Zeuzem S, Poordad F, Goodman ZD, Sings HL, Boparai N, Burroughs M, Brass CA, Albrecht JK, Esteban R; HCV RESPOND-2 Investigators. Boceprevir for previously treated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1207-17. doi: 10.1056/NEJMoa1009482. PMID 21449784

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 154 participants who discontinued during the treatment phase (including those from lead in and/or boceprevir/placebo) entered the follow up phase
Period: Treatment (Tx): 4 WEEK LEAD-IN PERIOD
Arm/Group | Placebo+PEG2b+RBV, x 44 Weeks | Boceprevir+PEG2b+RBV, Response Guided Therapy | Boceprevir+PEG2b+RBV, x 44 Weeks
Started | 80 | 162 | 162
Treated With PEG2b + RBV | 80 | 162 | 161
Completed | 78 | 156 | 160
Not Completed | 2 | 6 | 2
Not completed — Adverse Event | 1 | 3 | 1
Not completed — Subject withdrawal unrelated to Tx | 1 | 0 | 0
Not completed — Subject withdrawal related to Tx | 0 | 1 | 0
Not completed — Subject withdrew consent | 0 | 2 | 0
Not completed — Randomized but not treated | 0 | 0 | 1
Period: Tx: RECEIVING BOCEPREVIR/PLACEBO
Arm/Group | Placebo+PEG2b+RBV, x 44 Weeks | Boceprevir+PEG2b+RBV, Response Guided Therapy | Boceprevir+PEG2b+RBV, x 44 Weeks
Started | 78 | 156 | 160
Completed | 23 | 104 | 105
Not Completed | 55 | 52 | 55
Not completed — Adverse Event | 1 | 10 | 19
Not completed — Treatment Failure | 49 | 36 | 29
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Subject withdrawal unrelated to Tx | 3 | 1 | 4
Not completed — Subject withdrawal related to Tx | 2 | 0 | 1
Not completed — Subject withdrew consent | 0 | 2 | 1
Not completed — Non-compliance with protocol | 0 | 1 | 1
Not completed — Administrative | 0 | 1 | 0
Period: FOLLOWUP
Arm/Group | Placebo+PEG2b+RBV, x 44 Weeks | Boceprevir+PEG2b+RBV, Response Guided Therapy | Boceprevir+PEG2b+RBV, x 44 Weeks
Started | 77 | 151 | 158
Completed | 37 | 136 | 143
Not Completed | 40 | 15 | 15
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 6 | 4
Not completed — Subject withdrawal unrelated to Tx | 3 | 4 | 5
Not completed — Subject withdrew consent | 31 | 4 | 5
Not completed — Non-compliance with protocol | 5 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+PEG2b+RBV, x 44 Weeks | Boceprevir+PEG2b+RBV, Response Guided Therapy | Boceprevir+PEG2b+RBV, x 44 Weeks | Total
Number analyzed (Participants) | 80 | 162 | 161 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (8.1) | 52.9 (7.4) | 52.3 (7.7) | 52.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 64 | 49 | 135
  Male | 58 | 98 | 112 | 268

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR) Rate in the Full Analysis Set (FAS) Population.
Description: SVR is defined as undetectable plasma hepatitis C virus RNA (HCV-RNA) at Follow-up Week 24. This outcome measure evaluates SVR after treatment with boceprevir and PEG2b plus RBV versus PEG2b plus RBV alone in participants with chronic hepatitis C (CHC) genotype 1 who failed prior treatment.
Time Frame: At Follow-up Week 24
Population: FAS = all randomized subjects who received at least one dose of any study medication (Peg, RBV, or boceprevir/placebo).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo+PEG2b+RBV, x 44 Weeks | Boceprevir+PEG2b+RBV, Response Guided Therapy | Boceprevir+PEG2b+RBV, x 44 Weeks
Number analyzed (Participants) | 80 | 162 | 161
Percentage of Participants | 21.3 | 58.6 | 66.5
Statistical Analysis 1: Comparison: Placebo+PEG2b+RBV, x 44 Weeks vs Boceprevir+PEG2b+RBV, Response Guided Therapy; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Treatment Difference = 37.4, 95% CI [25.7 to 49.1] — Difference in percentage of participants who achieved SVR: experimental minus control
Statistical Analysis 2: Comparison: Placebo+PEG2b+RBV, x 44 Weeks vs Boceprevir+PEG2b+RBV, x 44 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Treatment Difference = 45.2, 95% CI [33.7 to 56.8] — Difference in percentage of participants who achieved SVR: experimental minus control

2. Secondary Outcome: Sustained Virologic Response (SVR) Rate in the Modified Intent to Treat (mITT) Population.
Description: SVR is defined as undetectable plasma HCV-RNA at Follow-up Week 24. This outcome measure evaluates SVR after treatment with boceprevir and PEG2b plus RBV versus PEG2b plus RBV alone in participants with CHC genotype 1 who failed prior treatment.
  This key secondary efficacy endpoint was added as per the second protocol amendment on 02 DEC 2009.
Time Frame: At Follow-up Week 24
Population: mITT = all randomized subjects who received at least one dose of boceprevir (experimental arms) or boceprevir placebo (control arm).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo+PEG2b+RBV, x 44 Weeks | Boceprevir+PEG2b+RBV, Response Guided Therapy | Boceprevir+PEG2b+RBV, x 44 Weeks
Number analyzed (Participants) | 78 | 156 | 160
Percentage of Participants | 21.8 | 60.9 | 66.9
Statistical Analysis 1: Comparison: Placebo+PEG2b+RBV, x 44 Weeks vs Boceprevir+PEG2b+RBV, Response Guided Therapy; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Treatment Difference = 39.1, 95% CI [27.2 to 51.0] — Difference in percentage of participants who achieved SVR: experimental minus control
Statistical Analysis 2: Comparison: Placebo+PEG2b+RBV, x 44 Weeks vs Boceprevir+PEG2b+RBV, x 44 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Treatment Difference = 45.1, 95% CI [33.4 to 56.8] — Difference in percentage of participants who achieved SVR: experimental minus control

3. Secondary Outcome: Number of Participants With Early Virologic Response.
Description: Having undetectable HCV-RNA at Week 2, 4, 8, or 12 was considered Early Virologic Response.
Time Frame: At Week 2, 4, 8, or 12
Population: FAS = all randomized subjects who received at least one dose of any study medication (Peg, RBV, or boceprevir/placebo).
Measure: Number; unit: participants
Arm/Group | Placebo+PEG2b+RBV, x 44 Weeks | Boceprevir+PEG2b+RBV, Response Guided Therapy | Boceprevir+PEG2b+RBV, x 44 Weeks
Number analyzed (Participants) | 80 | 162 | 161
participants
  Week 2 | 0 | 0 | 0
  Week 4 | 2 | 0 | 2
  Week 8 | 7 | 74 | 84
  Week 12 | 23 | 111 | 121

4. Secondary Outcome: Number of Participants With Undetectable HCV-RNA at Follow-up Week 12 and at 72 Weeks After Randomization.
Time Frame: At Follow-up Week 12 and at 72 weeks after randomization
Population: FAS = all randomized subjects who received at least one dose of any study medication (Peg, RBV, or boceprevir/placebo).
Measure: Number; unit: participants
Arm/Group | Placebo+PEG2b+RBV, x 44 Weeks | Boceprevir+PEG2b+RBV, Response Guided Therapy | Boceprevir+PEG2b+RBV, x 44 Weeks
Number analyzed (Participants) | 80 | 162 | 161
participants
  Follow-Up Week 12 | 16 | 97 | 105
  72 Weeks Post Randomization | 17 | 93 | 105

ADVERSE EVENTS:
Arm/Group | Placebo+PEG2b+RBV, x 44 Weeks | Boceprevir+PEG2b+RBV, Response Guided Therapy | Boceprevir+PEG2b+RBV, x 44 Weeks
Serious Adverse Events (participants affected / at risk) | 4/80 | 16/162 | 23/161
Other Adverse Events (participants affected / at risk) | 77/80 | 159/162 | 160/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+PEG2b+RBV, x 44 Weeks (N=80) | Boceprevir+PEG2b+RBV, Response Guided Therapy (N=162) | Boceprevir+PEG2b+RBV, x 44 Weeks (N=161)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOPERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS NECROTISING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PEPTIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 2 (3) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PARKINSONISM (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
HOMICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
PHLEBITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+PEG2b+RBV, x 44 Weeks (N=80) | Boceprevir+PEG2b+RBV, Response Guided Therapy (N=162) | Boceprevir+PEG2b+RBV, x 44 Weeks (N=161)
ANAEMIA (Blood and lymphatic system disorders) | 16 (20) | 70 (117) | 75 (125)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (3) | 4 (12) | 11 (18)
NEUTROPENIA (Blood and lymphatic system disorders) | 8 (12) | 23 (60) | 23 (43)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 10 (12)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 (8) | 4 (4) | 11 (12)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 14 (23) | 12 (16)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 15 (17) | 19 (22)
DIARRHOEA (Gastrointestinal disorders) | 13 (21) | 38 (59) | 40 (59)
DRY MOUTH (Gastrointestinal disorders) | 7 (8) | 21 (25) | 26 (32)
DYSPEPSIA (Gastrointestinal disorders) | 5 (5) | 11 (16) | 10 (13)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 9 (9) | 9 (9)
NAUSEA (Gastrointestinal disorders) | 30 (37) | 72 (89) | 68 (99)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 10 (11) | 5 (6)
VOMITING (Gastrointestinal disorders) | 6 (6) | 23 (27) | 24 (33)
ASTHENIA (General disorders) | 13 (20) | 30 (43) | 38 (59)
CHILLS (General disorders) | 24 (36) | 56 (94) | 50 (63)
FATIGUE (General disorders) | 40 (59) | 87 (137) | 92 (115)
INFLUENZA LIKE ILLNESS (General disorders) | 20 (20) | 41 (51) | 38 (44)
INJECTION SITE ERYTHEMA (General disorders) | 7 (17) | 22 (24) | 16 (33)
INJECTION SITE REACTION (General disorders) | 7 (10) | 9 (12) | 16 (17)
IRRITABILITY (General disorders) | 10 (13) | 31 (38) | 36 (41)
PAIN (General disorders) | 3 (5) | 11 (12) | 15 (15)
PYREXIA (General disorders) | 20 (32) | 45 (58) | 48 (67)
BRONCHITIS (Infections and infestations) | 6 (6) | 3 (5) | 6 (7)
NASOPHARYNGITIS (Infections and infestations) | 6 (9) | 5 (6) | 4 (4)
SINUSITIS (Infections and infestations) | 7 (7) | 7 (10) | 4 (5)
WEIGHT DECREASED (Investigations) | 7 (8) | 21 (27) | 15 (19)
DECREASED APPETITE (Metabolism and nutrition disorders) | 13 (15) | 37 (38) | 46 (56)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13 (15) | 34 (36) | 39 (53)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (7) | 13 (16) | 14 (15)
MYALGIA (Musculoskeletal and connective tissue disorders) | 19 (28) | 46 (82) | 35 (42)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4) | 10 (13)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 6 (7) | 11 (11) | 12 (17)
DIZZINESS (Nervous system disorders) | 8 (8) | 26 (29) | 26 (36)
DYSGEUSIA (Nervous system disorders) | 9 (9) | 70 (79) | 72 (86)
HEADACHE (Nervous system disorders) | 39 (50) | 69 (95) | 64 (82)
MEMORY IMPAIRMENT (Nervous system disorders) | 4 (5) | 10 (10) | 5 (5)
ANXIETY (Psychiatric disorders) | 6 (7) | 19 (25) | 20 (23)
DEPRESSION (Psychiatric disorders) | 12 (12) | 18 (21) | 28 (39)
INSOMNIA (Psychiatric disorders) | 19 (33) | 50 (65) | 47 (62)
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 (20) | 30 (36) | 40 (59)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 29 (42) | 40 (46)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 22 (23) | 14 (14)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (11) | 7 (9)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8) | 9 (9)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 11 (12)
ALOPECIA (Skin and subcutaneous tissue disorders) | 13 (14) | 42 (44) | 29 (30)
DRY SKIN (Skin and subcutaneous tissue disorders) | 7 (11) | 35 (40) | 37 (45)
PRURITUS (Skin and subcutaneous tissue disorders) | 14 (17) | 31 (41) | 31 (47)
RASH (Skin and subcutaneous tissue disorders) | 5 (6) | 27 (32) | 24 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may not publish/publicly present interim results without prior consent of Sponsor. Any materials that report results of the study must be sent to Sponsor 45 days prior to submission for publication/presentation. Sponsor has right to review and comment. In case of any disagreements concerning appropriateness of the materials, investigator and Sponsor must meet to make a good faith effort to discuss/resolve the issues or disagreement, prior to submission for publication/presentation.